CLINICAL TRIAL: NCT00570921
Title: A Phase II Study of Combined Fulvestrant (Faslodex) and Everolimus in Advanced/Metastatic Breast Cancer After Aromatase Inhibitor Failure
Brief Title: Study of Combined Fulvestrant and Everolimus in Advanced/Metastatic Breast Cancer After Aromatase Inhibitor Failure
Acronym: BRE-43
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mara Chambers (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Mara Chambers, Sponsor-Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-BRE-43-NP
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Results first posted 2014-12-31 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Fulvestrant; Everolimus
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fulvestrant + Everolimus (Experimental): Fulvestrant + Everolimus
  Fulvestrant was administered intramuscularly (in the gluteus maximus) in a loading dose schedule as follows: 500 mg in two divided doses-one on each side on day 1, then 250 mg on day 14, and then 250 mg on day 28 and every 4 weeks ± 3 days thereafter. Everolimus was administered initially at a dose of 5 mg daily in the first 5-patient cohort for the first month of treatment and then increased to 10 mg PO daily after that.
  Interventions: Drug: Everolimus; Drug: Fulvestrant

INTERVENTIONS:
Drug: Everolimus — Everolimus tablets, two-5 mg tablets a day
  Other Names: RAD001
Drug: Fulvestrant — intramuscular, 500 mg in two divided doses- one on each side- on day 1, then 250mg on day 14, then 250 mg on day 28 and every 4 weeks +/- 3 days thereafter
  Other Names: Faslodex

SUMMARY:
The primary objective of this study is to determine if estrogen receptor-targeted therapy with fulvestrant used in combination with Everolimus is an effective and safe therapy for women with hormone receptor positive metastatic breast cancer after failure of aromatase inhibitor therapy.

DETAILED DESCRIPTION:
Fulvestrant, which degrades ER, is used after aromatase inhibitor (AI) failure in metastatic breast cancer but resistance develops quickly. We hypothesized that using everolimus to inhibit mammalian target of rapamycin (mTOR), a key signaling pathway in endocrine resistance, may delay fulvestrant resistance in patients and thus improve its efficacy. We conducted a phase II trial of combined fulvestrant and everolimus in postmenopausal women with disease progression or relapse after an AI. Primary endpoint was time to progression (TTP) and secondary endpoints included objective response rate, clinical benefit rate (CBR), safety, and biomarker correlates. Tumor blocks were collected and biopsy of accessible tumor was done for future biomarker analysis.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal status, defined as any one of the following criteria: Documented history of bilateral oophorectomy, Age 60 years or more, OR Age 45 to 59 and satisfying one or more of the following criteria: Amenorrhea for at least 12 months and intact uterus OR Amenorrhea for less than 12 months and a follicle stimulating hormone (FSH) concentration - within postmenopausal range including: Patients who have had a hysterectomy or Patients who have received hormone replacement
* Patients must have histologically confirmed invasive breast cancer
* Metastatic or locally advanced disease
* Patients must have estrogen receptor and/or progesterone receptor positive disease
* Measurable or evaluable disease
* Failure of aromatase inhibitor therapy within the previous 6 months. Patients who received prior tamoxifen are eligible to enroll
* Prior aromatase inhibitor therapy or other endocrine therapy must be discontinued at least 1 week prior to enrollment and any toxicity from such therapy must have reverted to grade I or less at the time of enrollment
* Patients must not have received chemotherapy, radiation therapy, or had surgery within 4 weeks prior to enrollment and any toxicity from such therapy must have recovered to grade 1 or less prior to enrollment
* Patients must not have received either of the study medications previously
* WHO performance status of 0, 1, or 2
* Adequate organ function defined as follows: Adequate renal function, defined by a serum creatinine within the upper limits of normal, Adequate liver function, defined by a bilirubin of < 1.5 the upper limit of normal (ULN) and aspartate aminotransferase (AST), alanine aminotransferase (ALT) of ≤ 2.5 times the ULN, Adequate bone marrow function, defined as an absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelet count (PLT) >100,000/ul, Hb >9 gm/dl, international normalized ratio (INR) <1.3, and because fulvestrant is administered intramuscularly, it should not be used in patients with bleeding diatheses, thrombocytopenia or in patients on anticoagulants
* Patients will be asked to provide a tumor paraffin block if available
* Ability to understand and sign a written informed consent for participation in the trial

Exclusion Criteria:

* Known severe hypersensitivity to everolimus (or similar drugs) or any of the excipients of this product
* Premenopausal status
* Other coexisting malignancies with the exception of basal cell carcinoma or cervical cancer in situ
* Patients with brain metastasis or leptomeningeal involvement
* Patients with malignant pleural effusion or ascites only disease
* Rapidly progressive visceral disease
* WHO performance status of 3 or 4
* As judged by the investigator, uncontrolled intercurrent illness including, but not limited to: Ongoing or active infection, Symptomatic congestive heart failure, Unstable angina pectoris or significant cardiac arrhythmia, Psychiatric illness/social situations that would limit compliance with study requirements, Severely impaired lung function such as severe chronic obstructive pulmonary disease (COPD) or interstitial lung disease, a known forced expiratory volume at one second (FEV1) of < 1.5 liters, or dyspnea of grade III or greater, Uncontrolled diabetes as defined by a fasting blood sugar (FBS) of > 1.5 ULM, Known liver disease such as cirrhosis or chronic hepatitis, Known HIV positivity, OR known condition causing malabsorption
* Chronic treatment with systemic steroids or other immunosuppressive agents
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the clinical trial
* Prior treatment with an mTOR inhibitor
* Treatment with a non-approved or investigational drug within 30 days or 5 half-lives of the drug, whichever is greater, before Day 1 of study treatment
* In the opinion of the investigator, bleeding diathesis or anticoagulation therapy that would preclude intramuscular injections
* History of hypersensitivity to castor oil

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-04; Primary Completion 2013-02 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mara Chambers, M.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

REFERENCES:
- [Result] Massarweh S, Romond E, Black EP, Van Meter E, Shelton B, Kadamyan-Melkumian V, Stevens M, Elledge R. A phase II study of combined fulvestrant and everolimus in patients with metastatic estrogen receptor (ER)-positive breast cancer after aromatase inhibitor (AI) failure. Breast Cancer Res Treat. 2014 Jan;143(2):325-32. doi: 10.1007/s10549-013-2810-9. Epub 2013 Dec 11. PMID 24327334

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at a single location, University of Kentucky Markey Cancer Center, between March 2008 and October 2012.
Period: Overall Study
Arm/Group | Fulvestrant + Everolimus
Started | 33
Completed | 31
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: 2 were not evaluable as described in participant flow and not included in demographic table.
Groups:
- Fulvestrant & Everolimus: Fulvestrant + Everolimus
  Fulvestrant was administered intramuscularly (in the gluteus maximus) in a loading dose schedule as follows: 500 mg in two divided doses-one on each side on day 1, then 250 mg on day 14, and then 250 mg on day 28 and every 4 weeks ± 3 days thereafter. Everolimus was administered initially at a dose of 5 mg daily in the first 5-patient cohort for the first month of treatment and then increased to 10 mg PO daily after that.
  Everolimus: Everolimus tablets, two-5 mg tablets a day
  Fulvestrant: intramuscular, 500 mg in two divided doses- one on each side- on day 1, then 250mg on day 14, then 250 mg on day 28 and every 4 weeks +/- 3 days thereafter
Arm/Group | Fulvestrant & Everolimus
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: years] | 54 [45 to 85]
Gender [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 27
  Black | 3
  Hispanic | 1
Hormone Receptor Status [Number; unit: participants]
  ER-positive/progesterone receptor (PgR)-positive | 26
  ER-positive/progesterone receptor (PgR)-negative | 5
Human epidermal growth factor receptor 2 (HER2) Status [Number; unit: participants]
  Negative | 29
  Positive | 2
Histology [Number; unit: participants]
  Ductal | 26
  Lobular | 3
  Mixed ductal and lobular | 1
  Intracystic papillary | 1
Relapsed versus de novo metastasis [Number; unit: participants]
  Relapse | 24
  De novo | 7
Number of metastatic sites [Number; unit: participants]
  1 | 4
  2 | 10
  3 or more | 17
Bone Disease [Number; unit: participants]
  Yes | 20
  No | 11
Liver Disease [Number; unit: participants]
  Yes | 19
  No | 12
Lung Disease [Number; unit: participants]
  Yes | 17
  No | 14
Intact Primary Tumor [Number; unit: participants]
  Yes | 6
  No | 25
Skin Disease [Number; unit: participants]
  Yes | 4
  No | 27
Prior aromatase inhibitor (AI) therapy within 6 months of enrollment [Number; unit: participants] | 31
Prior tamoxifen therapy [Number; unit: participants]
  Yes | 25
  No | 6
Prior Chemotherapy [Number; unit: participants]
  Yes | 22
  No | 9
3 or more prior endocrine therapies [Number; unit: participants]
  Yes | 8
  No | 23
Two prior aromatase inhibitor therapy [Number; unit: participants]
  Yes | 7
  No | 24
AI Sensitivity [Number; unit: participants]
  Sensitive | 21
  Resistant | 10

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Time Frame: Duration of time start of treatment to time of documented progression or death
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fulvestrant + Everolimus
Number analyzed (Participants) | 31
months | 7.4 [1.9 to 12.1]
Statistical Analysis 1: Comparison: Fulvestrant + Everolimus; We hypothesized that median time to progression (TTP) in our trial will increase from 3.7 months for the historical fulvestrant-only control to 7.0 months on the combination of fulvestrant and everolimus in the current trial. A sample of 40 evaluable patients was calculated to show the increase in TTP with 80% power and 5% significance level based on a two sided test of differences in survival times between historical controls and treated group; Test type: Superiority or Other; Median Time to Progression = 7.4, 95% CI 2-sided [1.9 to 12.1]

2. Secondary Outcome: Objective Response Rates
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Evaluated 60 days after therapy start
Measure: Number; unit: participants
Arm/Group | Fulvestrant + Everolimus
Number analyzed (Participants) | 31
participants | 4
Statistical Analysis 1: Comparison: Fulvestrant + Everolimus; Test type: Superiority or Other; Response Rate Percentage = 12.9, 95% CI 2-sided [3.63 to 29.83] — Percentage of Patients with a complete or partial response with 95% exact binomial proportion confidence interval

3. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate is defined as a complete response, partial response, or stable disease (CR, PR, SD) by Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for a minimum of at least 24 weeks or more.
Time Frame: Duration of response or stable disease for 24 weeks or more
Measure: Number; unit: participants
Arm/Group | Fulvestrant + Everolimus
Number analyzed (Participants) | 31
participants | 15
Statistical Analysis 1: Comparison: Fulvestrant + Everolimus; Test type: Superiority or Other; Percentage with clinical benefit = 48.39, 95% CI 2-sided [30.15 to 66.94] — Percentage of patients that had a complete response, partial response, or stable disease for 24 weeks or more as defined by RECIST v1.0

ADVERSE EVENTS:
Arm/Group | Fulvestrant + Everolimus
Serious Adverse Events (participants affected / at risk) | 5/33
Other Adverse Events (participants affected / at risk) | 31/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant + Everolimus (N=33)
Left Ventricular Thrombus (Cardiac disorders) | 1
Acute Cholecystitis (Hepatobiliary disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant + Everolimus (N=33)
AST Elevation (Investigations) | 27
ALT Elevation (Investigations) | 24
Anemia (Blood and lymphatic system disorders) | 23
Hyperglycemia (Metabolism and nutrition disorders) | 22
Hypercholesterolemia (Investigations) | 21
Hypokalemia (Metabolism and nutrition disorders) | 19
Mucositis (Respiratory, thoracic and mediastinal disorders) | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 17
Hypoalbuminemia (Metabolism and nutrition disorders) | 17
Weight loss (Investigations) | 15
Leukopenia (Blood and lymphatic system disorders) | 14
Rash/skin changes (Skin and subcutaneous tissue disorders) | 13
Nausea (Gastrointestinal disorders) | 10
Fatigue (General disorders) | 10
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 6
Edema (General disorders) | 6
Joint pain (Musculoskeletal and connective tissue disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 6
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 5
Itching/dry skin only (Skin and subcutaneous tissue disorders) | 3

LIMITATIONS AND CAVEATS:
Potential toxicities of mammalian target of rapamycin (mTOR) inhibitors and our observation that a third of patients had no benefit from this strategy, we need to identify biomarkers that correlate with treatment benefit for better patient selection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No